CLINICAL TRIAL: NCT04663295
Title: Safety, Effectiveness and Usability Evaluation of the Hybrid Closed Loop (HCL) System in Type 1 Adult and Adolescent Subjects in Chinese Population
Brief Title: MiniMed™ 670G System China Study for Type I Diabetic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP329
Record Dates: First submitted 2020-10-28; First posted 2020-12-11 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects with Type 1 diabetes wearing HCL pump system (Experimental): Subjects 14-75 years of age who have been diagnosed with Type 1 diabetes.
  Interventions: Device: MiniMed™ 670G system

INTERVENTIONS:
Device: MiniMed™ 670G system — Hybrid closed loop insulin pump with associated CGM and blood glucose meter

SUMMARY:
The purpose of this study is to obtain clinical data in Chinese patients to support product registration of the MiniMed™ 670G system with the National Medical Product Administration (NMPA) in China. The results from the study will be submitted to the NMPA for product registration.

DETAILED DESCRIPTION:
This study is a multi-center, single arm study in insulin-requiring subjects with type 1 diabetes who are 14 years of age and older. The run-in period will be approximately up to 35 days long, followed by a study period that will be approximately up to 33 days in duration.

The study is anticipated to last no longer than 13 months from investigational center initiation to completion of all data entry and monitoring procedures. The study will target approximately 5 months to complete subject enrollment. Subjects can expect to participate for approximately 2-3 months including the run-in and study periods.

A total of up to 75 subjects (aged 14-75) will be enrolled at a minimum 2 investigational centers and up to 6 investigational centers (hospitals) in China to have at least 50 subjects who complete the study.

The MiniMed™ HCL system that was employed in this study was the MiniMed™ 670G Bluetooth version (MMT-1883). The MiniMed™ 670G system with Bluetooth™ technology is the MiniMed™ 770G system.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is age 14- 75 years at time of Screening.
2. Subject has a clinical diagnosis of type 1 diabetes for 2 years or more as determined via medical record or source documentation by an individual qualified to make a medical diagnosis.

   Study-specific inclusion criteria
3. Subject is willing to perform ≥ 4 finger stick BG measurements daily.
4. Subject is willing to perform required sensor calibrations.
5. Subject is willing to wear the system continuously throughout the study.
6. Subject must have a minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units.
7. Subject has a Glycosylated hemoglobin (HbA1c) less than 10% (as processed by the investigational center lab or their contracted Local Lab) at time of Screening visit.
8. Subject has thyroid-stimulating hormone (TSH) in the normal range OR if the TSH is out of normal reference range the Free T3 is below or within the lab's reference range and Free T4 is within the normal reference range. Prior labs in the last 6 months are sufficient.
9. Subject has been on pump therapy for greater than 6 months prior to screening (with or without CGM experience).
10. Subject is willing to upload data from the study pump and meter at home.
11. If subject has celiac disease, it has been adequately treated as determined by the investigator.
12. Subject has been taking and is willing to take one of the following insulins throughout the course of the study:

    * Humalog™* (insulin lispro injection)
    * NovoLog™* (insulin aspart)
13. Subject must be able to carbohydrate count or willing to learn how to carbohydrate count for the study.

Exclusion Criteria:

1. Subject has a history of 2 or more episodes of severe hypoglycemia, which resulted in any the following during the 6 months prior to Screening:

   1. Medical assistance (i.e. Paramedics, Emergency Room (ER) or Hospitalization)
   2. Coma
   3. Seizures
2. Subject has been hospitalized or has visited the ER in the 6 months prior to Screening resulting in a primary diagnosis of uncontrolled diabetes.
3. Subject has had DKA in the 6 months prior to Screening.
4. Subject is unable to tolerate tape adhesive in the area of sensor placement.
5. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
6. Subject is a female of child-bearing potential who has a positive pregnancy test at Screening or plans to become pregnant during the course of the study.
7. Subject is a female who is sexually active and able to conceive should be excluded if they are not using an effective method of contraception and do not agree to continue using an effective method of contraception for the duration of the study as determined by investigator.
8. Subject has had any of the following cardiovascular events within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease.
9. Subject is being treated for hyperthyroidism at time of Screening.
10. Subject has a diagnosis of adrenal insufficiency.
11. Subject has taken any oral, injectable, or intravenous (IV) glucocorticoids within 8 weeks from time of Screening, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
12. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks. (Please note participation in an observational study is acceptable.)
13. Subject is currently abusing illicit drugs.
14. Subject is currently abusing alcohol.
15. Subject is using pramlintide (Symlin), DPP-4 inhibitor, liraglutide (Victoza or other GLP-1 agonists), metformin, canagliflozin (Invokana or other SGLT2 inhibitors) at time of Screening.
16. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator.
17. Subject has elective surgery planned that requires general anesthesia during the course of the study.
18. Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of Screening
19. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
20. Subject diagnosed with current eating disorder such as anorexia or bulimia
21. Subject has been diagnosed with chronic kidney disease that results in chronic anemia.
22. Subject has a hematocrit (Hct) that is below the normal reference range of lab used. Prior labs in the last 6 months are sufficient.
23. Subject is on dialysis.
24. Subject has an estimated glomerular filtration rate (eGFR) of < 30.
25. Subject has a pediatric BMI category of underweight (less than the 5th percentile) as defined by Centers for Disease Control (CDC) (https://www.cdc.gov/healthyweight/assessing/bmi/childrens_bmi/about_childrens_bmi.html)
26. Subject is a member the research staff involved with the study.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Mu, MD, Principal Investigator — Chinese PLA General Hospital; Yan Bi, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Yongde Peng, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Yanbing Li, MD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (4):
- China (4):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Shanghai General Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pei Y, Ke W, Lu J, Lin Y, Zhang Z, Peng Y, Bi Y, Li Y, Hou J, Zhang X, Chen X, Treminio Y, Lee SW, Shin J, Rhinehart AS, Vigersky RA, Mu Y. Safety Event Outcomes and Glycemic Control with a Hybrid Closed-Loop System Used by Chinese Adolescents and Adults with Type 1 Diabetes Mellitus. Diabetes Technol Ther. 2023 Oct;25(10):718-725. doi: 10.1089/dia.2023.0234. Epub 2023 Sep 5. PMID 37578804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started on 31Oct2020 and ended on 30Apr2021. Recruitment was conducted at four hospitals.
Pre-assignment Details: There were 74 participants screened in the study. Of the 74 participants, 8 participants failed screening, and 1 participant was withdrawn prior to run-in. Therefore, 65 participants started run-in period. A total of 3 participants were withdrawn during the run-in period. Therefore, a total of 62 participants were included in the Intention to Treat Population and started the study period.
Groups:
- Participants With Type 1 Diabetes Wearing HCL Pump System: Participants 14-75 years of age who have been diagnosed with Type 1 diabetes and wore MiniMed™ 670G system.
Period: Run-in Period
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Started | 65
Completed | 62
Not Completed | 3
Not completed — Withdrawal by Subject | 3
Period: Overall Study Period
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Started | 62
Completed | 60
Not Completed | 2
Not completed — Pregnancy | 1
Not completed — Withdrawn by Parent/Guardian | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat Population.
Groups:
- Participants With Type 1 Diabetes Wearing HCL Pump System: Participants 14-75 years of age who have been diagnosed with Type 1 diabetes and wore MiniMed™ 670G system during study period.
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han Chinese | 62
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.1 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Time in Target Range (% of Sensor Glucose (SG)): 70 mg/dL (3.9 mmol/L) ≤ SG ≤ 180 mg/dL (10 mmol/L)
Description: The overall mean change in % of time in target range from run-in period to study period will be estimated and compared by a simple superiority paired test and a significance level of 0.025 (one-sided).
Time Frame: Baseline to end of 1-month study
Population: Intention to Treat Population.
Measure: Mean (Standard Deviation); unit: percentage of total readings
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
percentage of total readings
  Baseline | 75.3 (12.4)
  1-month Study | 80.9 (7.5)
  Change | 5.6 (9.1)
Statistical Analysis 1: Comparison: Participants With Type 1 Diabetes Wearing HCL Pump System; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney) — One-sided test at significant level of 0.025; Wilcoxon Signed rank test comparing baseline and study period; Mean Difference (Net) = 5.6, 95% CI 2-sided [3.3 to 7.9]

2. Secondary Outcome: Time in Hypoglycemic Range
Description: Time in hypoglycemic range (% of SG): SG < 70 mg/dL (3.9 mmol/L), SG < 60 mg/dL (3.3 mmol/L), SG < 54 mg/dL (3.0 mmol/L) will be summarized.
Time Frame: 1-month study
Population: Intention to Treat Population
Measure: Mean (Standard Deviation); unit: percentage of total readings
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
percentage of total readings
  SG < 54 mg/dL (3.0 mmol/L) | 0.4 (0.4)
  SG < 60 mg/dL (3.3 mmol/L) | 0.8 (0.7)
  SG < 70 mg/dL (3.9 mmol/L) | 2.2 (1.5)

3. Secondary Outcome: Time in Hyperglycemic Range: SG > 180 mg/dL (10 mmol/L), 250 mg/dL (13.9 mmol/L) and 350 mg/dL (19.4 mmol/L)
Description: Time in hyperglycemic range (SG > 180 mg/dL (10 mmol/L), 250 mg/dL (13.9 mmol/L) and 350 mg/dL (19.4 mmol/L)) will be summarized.
Time Frame: 1-month study
Population: Intention to Treat Population.
Measure: Mean (Standard Deviation); unit: percentage of total readings
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
percentage of total readings
  SG > 180 mg/dL (10 mmol/L) | 16.9 (7.5)
  SG > 250 mg/dL (13.9 mmol/L) | 2.4 (2.4)
  SG > 350 mg/dL (19.4 mmol/L) | 0.1 (0.2)

4. Secondary Outcome: Standard Deviation (SD) of SG in mmol/L
Description: In order to evaluate glucose variation, we calculated standard deviation. The standard deviation (SD) of SG will be summarized in the unit of mmol/L
Time Frame: 1-month study
Population: Intention to Treat Population.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
mmol/L | 2.4 (0.4)

5. Secondary Outcome: Standard Deviation (SD) of SG in mg/dL
Description: In order to evaluate glucose variation, we calculated standard deviation. The standard deviation (SD) of SG will be summarized in the unit of mg/dL.
Time Frame: 1-month study
Population: Intention to Treatment Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
mg/dL | 43.2 (7.8)

6. Secondary Outcome: Coefficient of Variation (CV) of SG
Description: In order to evaluate glucose variation, we calculated coefficient of variation (CV) of SG. The glucose coefficient of variation (CV) will be summarized in percentage.
Time Frame: 1-month study
Population: Intention to Treat Population.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
Percentage | 30.6 (4.2)

7. Secondary Outcome: Change of Total Daily Dose (TDD) of Insulin From Baseline to End of Study (EOS)
Description: Change of Total Daily Dose (TDD) of insulin from baseline to EOS will be summarized.
Time Frame: Baseline to end of 1-month study
Population: Intention to Treat Population.
Measure: Mean (Standard Deviation); unit: Units/Day
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
Units/Day
  Baseline | 42.8 (19.8)
  End of 1-month study | 40.7 (18.9)
  Change | -2.1 (9.8)

8. Secondary Outcome: Change of Weight From Baseline to EOS
Description: Change of weight from baseline to EOS will be summarized.
Time Frame: Baseline to end of 1-month study
Population: Intention to Treat Population with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 60
Kg
  Baseline | 61.0 (10.5)
  End of 1-month study | 61.0 (10.1)
  Change | 0.1 (1.9)

9. Secondary Outcome: Time Spent in Auto Mode (HCL) Versus Time Spent in Manual Mode (Open Loop)
Description: Time spent in Auto Mode (HCL) and time spent in Manual Mode (open loop) will be summarized.
Time Frame: 1-month study
Population: Intention to Treat Population.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Participants With Type 1 Diabetes Wearing HCL Pump System
Number analyzed (Participants) | 62
percentage of time
  Time spent in Auto Mode | 93.5 (8.2)
  Time spent in Manual Mode | 6.5 (8.2)

10. Secondary Outcome: Time in Specific Range Stratified by Baseline HbA1c Ranges (< 7%, 7 - < 7.5%, 7.5 - 8%, > 8%)
Description: Time in target range (% of SG): 70 mg/dL (3.9 mmol/L) ≤ SG ≤ 180 mg/dL (10 mmol/L) in study period Time in hypoglycemic range (% of SG): SG < 70 mg/dL (3.9 mmol/L), 60 mg/dL (3.3 mmol/L) and 54 mg/dL (3.0 mmol/L) in study period Time in hyperglycemic range: SG > 180 mg/dL (10 mmol/L), 250 mg/dL (13.9 mmol/L) and 350 mg/dL (19.4 mmol/L) in study period
Time Frame: 1-month study
Population: Intention to Treat Population at each subgroup.
Measure: Mean (Standard Deviation); unit: percentage of total readings
Groups:
- Participants With Baseline HbA1c < 7%: Participants 14-75 years of age with baseline HbA1c < 7%, who have been diagnosed with Type 1 diabetes and wore MiniMed™ 670G system during study period.
- Participants With Baseline 7% ≤ HbA1c < 7.5%: Participants 14-75 years of age with baseline HbA1c < 7.5% and ≥ 7%, who have been diagnosed with Type 1 diabetes and wore MiniMed™ 670G system during study period.
- Participants With Baseline 7.5% ≤ HbA1c ≤ 8.0%: Participants 14-75 years of age with baseline HbA1c ≤ 8% and ≥ 7.5%, who have been diagnosed with Type 1 diabetes and wore MiniMed™ 670G system during study period.
- Participants With Baseline HbA1c > 8.0%: Participants 14-75 years of age with baseline HbA1c > 8%, who have been diagnosed with Type 1 diabetes and wore MiniMed™ 670G system during study period.
Arm/Group | Participants With Baseline HbA1c < 7% | Participants With Baseline 7% ≤ HbA1c < 7.5% | Participants With Baseline 7.5% ≤ HbA1c ≤ 8.0% | Participants With Baseline HbA1c > 8.0%
Number analyzed (Participants) | 29 | 12 | 11 | 10
percentage of total readings
  SG < 54 mg/dL (3.0 mmol/L) | 0.3 (0.3) | 0.4 (0.4) | 0.4 (0.3) | 0.6 (0.6)
  SG < 60 mg/dL (3.3 mmol/L) | 0.7 (0.6) | 0.8 (0.7) | 0.9 (0.4) | 1.3 (1.0)
  SG < 70 mg/dL (3.9 mmol/L) | 2.0 (1.4) | 2.0 (1.4) | 2.2 (0.8) | 3.1 (2.1)
  70 mg/dL (3.9 mmol/L) ≤ SG ≤ 180 mg/dL (10 mmol/L) | 85.1 (5.6) | 78.1 (5.6) | 80.0 (5.2) | 72.8 (8.6)
  SG > 180 mg/dL (10 mmol/L) | 12.9 (5.4) | 19.9 (5.4) | 17.9 (5.1) | 24.1 (9.8)
  SG > 250 mg/dL (13.9 mmol/L) | 1.2 (1.1) | 2.9 (1.9) | 2.6 (1.5) | 4.9 (3.9)
  SG > 350 mg/dL (19.4 mmol/L) | 0.0 (0.1) | 0.1 (0.2) | 0.1 (0.1) | 0.3 (0.3)

ADVERSE EVENTS:
Time Frame: 2-4 weeks run in period and 1-month study period
Description: AE events prior run-in were not reported in this section.
Groups:
- Subjects With Type 1 Diabetes Wearing HCL Pump System During Run in Period: Subjects 14-75 years of age who have been diagnosed with Type 1 diabetes and wore MiniMed™ 670G system during Run in period.
- Subjects With Type 1 Diabetes Wearing HCL Pump System During Study Period: Subjects 14-75 years of age who have been diagnosed with Type 1 diabetes and wore MiniMed™ 670G system during study period.
Arm/Group | Subjects With Type 1 Diabetes Wearing HCL Pump System During Run in Period | Subjects With Type 1 Diabetes Wearing HCL Pump System During Study Period
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/62
Other Adverse Events (participants affected / at risk) | 6/65 | 9/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Type 1 Diabetes Wearing HCL Pump System During Run in Period (N=65) | Subjects With Type 1 Diabetes Wearing HCL Pump System During Study Period (N=62)
Infusion site haemorrhage (General disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4)
Diabetic ketosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) — For study period, one is device related, the other is non-device related.
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) — For run in period: One is device Device related severe hyperglycemia, the other is not device related. For study period: Device related severe hyperglycemia.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT04663295/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT04663295/SAP_001.pdf